CLINICAL TRIAL: NCT06532266
Title: A Randomised Controlled Trial Using Active Warming in Prevention of Newborn Hypothermia After Caesarean Delivery Without Interruption to Skin-to-skin Contact
Brief Title: Randomised Controlled Trial on Using Active Warming to Prevent Newborn Hypothermia After Caesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW 22-695
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Newborn; Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Device: TechTrade Ready Heat Half Body Temperature Management Blankets
- Control (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Device: TechTrade Ready Heat Half Body Temperature Management Blankets — The thermal blanket will be placed on top of the cotton blanket. Newborn will be first covered with conventional warm blanket then adding the thermal blanket on top. The thermal blanket will be placed inside a "pillowcase" like cotton blanket to avoid direct contact with mother or newborn.
  Arms: Intervention
Other: Control — 3 layers of 100% cotton woven blankets
  Arms: Control

SUMMARY:
Despite the enormous advantages that skin-to-skin contact (STSC) and Delaying Cord Clamping (DCC) bring, newborns can lose heat quickly if they are not thermally protected. In the first 10-20 minutes after birth, newborns can experience a body temperature drop of between 2°C to 4°C if they are not properly dried and covered. In 2014, Horn et al. published a research paper regarding the incidence and prevention of newborn hypothermia after Caesarean delivery. The findings showed up to 80% of newborns become hypothermic if only warm towels (passive insulation) were used during STSC after Caesarean delivery. Evidence also shows higher hypothermia rates in infants born by Caesarean section than vaginal birth.

STSC will begin while Caesarean section continues. Newborns will be clothed in a cotton hat and diaper. Newborns will be placed on bare chest of mother, horizontally, in prone position. The head of the newborn will turn laterally, making the nose and mouth unobstructed. Newborns' hands are not swaddled and are free to move to allow exploration to facilitate first feeding. In both groups, infants will be covered from head-to-toe with 3 layers of 100% cotton woven blankets, taken from a 70°C heating cabinet. For the "intervention group", thermal blanket will be placed on top of the cotton blanket. Newborn will be first covered with conventional warm blanket then adding the thermal blanket on top. The thermal blanket will be placed inside a "pillowcase" like cotton blanket to avoid direct contact with mother or newborn.

ELIGIBILITY:
Inclusion Criteria:

* All women scheduled for elective Caesarean section under spinal anaesthesia during study period.

Exclusion Criteria:

* Multiple pregnancy
* Gestation <37week or >42 week
* Placenta previa or abruptio placenta
* Abnormal Cardiotocogram or fetal heart rate immediately prior to Caesarean section
* Suspected or known fetal congenital abnormality
* Immediate newborn condition that prevents STSC

  * Newborn birth weight <2.5kg
  * Newborn rectal temperature >38°C
  * Maternal tympanic temperature >38°C

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Newborn hypothermia | after 20 minutes of skin to skin contact after Caesarean delivery or at the cessation of using active or conventional warming method before completion of 20 minutes of STSC, whichever happens first.
  Body temperature below 36.5°C

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wang Cheung, MD, Study Director — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided